CLINICAL TRIAL: NCT03890731
Title: A Single Arm, Open-label, Multicenter Phase 2 Study of Regorafenib in Participants Who Have Been Treated in a Previous Bayer-sponsored Regorafenib Study (Monotherapy or Combination Treatment) That Has Reached the Primary Completion Endpoint or the Main Data Analysis, or Has Been Stopped Prematurely.
Brief Title: A Clinical Study of Regorafenib in Participants Who Have Been Treated in Previous Bayer-sponsored Regorafenib Studies That Have Been Completed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20328; 2018-003650-24 (EudraCT Number)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Solid Cancer
Keywords: Metastatic colorectal cancer (mCRC); Renal cell cancer; Gastro-intestinal stromal tumor; Hepatocellular carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Renal Cell; Carcinoma, Hepatocellular | interventions — regorafenib; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patients (Other): Adult patients from completed Bayer-sponsored regorafenib trials who are benefitting from regorafenib treatment.
  Interventions: Drug: BAY73-4506 (Regorafenib, Stivarga)

INTERVENTIONS:
Drug: BAY73-4506 (Regorafenib, Stivarga) — Regorafenib is administered orally as 20 or 40 mg tablets at the dose that each patient received during the last cycle of the feeder trial. The dose may be either 60, 80, 120 or 160 mg once daily for 3 weeks of every 4-week cycle (3 weeks on, 1 week off).
  Other Names: Tyrosine-kinase inhibitor

SUMMARY:
The purpose of this study is to enable participants, currently receiving regorafenib in a Bayer-sponsored clinical trial, to continue treatment after their respective study has been closed. Patients participating in this study will be observed to collect information on how safe the drugs are and how this treatment is tolerated.

DETAILED DESCRIPTION:
The primary objectives of the study are a) to allow patients from Bayer-sponsored trials to continue regorafenib treatment after their respective study has been completed, and b) to further assess the safety of regorafenib. Secondary objective is the documentation of drug tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be age-eligible in the feeder study at the time of signing the informed consent.
* Participant is currently participating in any Bayer-sponsored regorafenib study and is receiving study treatment.
* Participant is currently benefiting from treatment with regorafenib monotherapy and meets criteria to initiate a subsequent cycle of therapy, as determined by the guidelines of the feeder protocol.
* Any ongoing adverse events that require temporary treatment interruption must be resolved to baseline grade or assessed as stable and not requiring further treatment interruption by the investigator.

Exclusion Criteria:

* Medical reasons not to start the next treatment cycle in the respective feeder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Tampa General Medical Group, Tampa, Florida, United States
- Germany (2):
  - Eberhard-Karls-Universität Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
- A.O.U. Careggi, Florence, Tuscany, Italy
- Saiseikai Utsunomiya Hospital, Utsunomiya, Tochigi, Japan
- Mount Vernon Hospital, Northwood, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/20328
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in multiple centers located in 5 countries (including Germany, Japan, Italy, United Kingdom, United States), first subject first visit of the study was on 02 APR 2019 and last subject last visit was on 28 FEB 2023.
Pre-assignment Details: This was a rollover study designed to enroll participants from ongoing or future feeder studies. Overall, 6 subjects were enrolled and treated in this study.
Groups:
- Regorafenib: Adult patients from completed Bayer-sponsored regorafenib trials who were benefitting from regorafenib treatment.
Period: Overall Study
Arm/Group | Regorafenib
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progressive disease | 1
Not completed — Patient's decision | 1
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An SAE was defined as any untoward medical occurrence that, at any dose: 1. results in death 2. is life-threatening 3. requires inpatient hospitalization or prolongation of existing hospitalization, etc.
Time Frame: from the signing of the informed consent form (ICF) until the safety follow up-visit (a duration of approximately 46 months)
Population: SAF
Measure: Number; unit: participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 6
participants
  Any AE | 6
  - Non-serious | 6
  - Serious | 3

2. Primary Outcome: Severity (by Worst Grade) of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: AEs were categorized by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: as for outcome 1
Population: SAF
Measure: Number; unit: participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 6
participants
  Worst grade - Grade 1 | 0
  Worst grade - Grade 2 | 2
  Worst grade - Grade 3 | 1
  Worst grade - Grade 4 | 3
  Worst grade - Grade 5 (death) | 0

3. Primary Outcome: Number and Severity of Participants With Drug-related Adverse Events (AEs) and Serious AEs (SAEs)
Description: A drug-related adverse event was any AE judged by investigator as having a reasonable suspected causal relationship to study drug.
Time Frame: as for outcome 1
Population: SAF
Measure: Number; unit: participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 6
participants
  Any AE | 5
  - Non-serious | 5
  - Serious | 1

4. Primary Outcome: Severity (by Worst Grade) of Participants With Drug-related Adverse Events (AEs) and Serious AEs (SAEs)
Description: A drug-related adverse event was any AE judged by investigator as having a reasonable suspected causal relationship to study drug.
  AEs were categorized by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: as for outcome 1
Population: SAF
Measure: Number; unit: participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 6
participants
  Worst grade - Grade 1 | 1
  Worst grade - Grade 2 | 3
  Worst grade - Grade 3 | 0
  Worst grade - Grade 4 | 1
  Worst grade - Grade 5 (death) | 0

5. Secondary Outcome: Number of Participants With Dose Modifications
Time Frame: as for outcome 1
Population: SAF
Measure: Number; unit: participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 6
participants
  Any modification | 6
  Interruption/Delay | 2
  Drug withdrawn | 5

ADVERSE EVENTS:
Time Frame: from the signing of the informed consent form (ICF) until the safety follow up-visit (a duration of approximately 46 months)
Description: The study had no dosage arms/groups as it was a rollover study.
Groups:
- Regorafenib: Adult patients from completed Bayer-sponsored regorafenib trials who are benefitting from regorafenib treatment.
Arm/Group | Regorafenib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (N=6)
Peritonitis (Infections and infestations) | 1 (1)
Electrocardiogram change (Investigations) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (3)
Retinal vein occlusion (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (11)
International normalised ratio increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (3)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (4)
Hypertension (Vascular disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03890731/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT03890731/SAP_001.pdf